CLINICAL TRIAL: NCT04065594
Title: Platelet Rich Plasma (PRP) Bio Stimulant Gel Dressing in Treating Chronic Non Healing Leg and Foot Ulcers: Cost and Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, clinical professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: zagazig university 1
Record Dates: First submitted 2019-08-12; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Ulcer Foot; Chronic Skin Ulcer; Non-Healing Ulcer of Skin
Keywords: ulcers; platelet rich plasma; ordinary dressing; non-healing
MeSH Terms: conditions — Foot Ulcer; Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP dressing (Experimental)
  Interventions: Procedure: PRP dressing
- conventional ordinary dressing (Experimental)
  Interventions: Procedure: conventional ordinary dressing

INTERVENTIONS:
Procedure: PRP dressing — PRP dressing gel dressings for treatment of chronic ulcer
  Arms: PRP dressing
Procedure: conventional ordinary dressing — conventional ordinary dressing for treatment of chronic ulcer
  Arms: conventional ordinary dressing

SUMMARY:
Background

Chronic non-healing ulcer is a common problem met in clinical practice and represents a burden to the patients. Chronic ulcer lacks growth factors (GFs) to promote the healing process and is frequently followed by superadded infections. Ordinary technique such as wound debridement and regular dressings cannot provide adequate results as these techniques cannot provide the necessary GFs. Platelet-rich plasma (PRP) helps wound healing by releasing various types of GFs.

The aim: to evaluate and compare the efficacy of PRP dressing versus traditional dressings in the treatment of chronic non-healing leg and foot ulcers of different etiology as regard cost of overall treatment and effectiveness (reduction of the size of the ulcer and safety of the technique).

Methods

This prospective study was performed on inpatients and outpatients in general surgery department, Zagazig university hospital from June 2017 to January 2019. Patients were divided randomly into two groups: group A received PRP dressing (N=22, 50%) and group B received conventional ordinary dressing (N=22, 50%).The mean follow-up period was 3 months after the last dressing. Patients treated with PRP at once-weekly interval for a maximum of 12 dressings while patients with ordinary dressings may need one dressing every other day for a maximum of 12 weeks. The reduction in the size of the ulcers (area and volume) in both groups was assessed using centimeter scale and Digital photographs before and after each session and during follow up period.

Keywords: Platelet-rich plasma, ulcers, non-healing, ordinary dressing.

DETAILED DESCRIPTION:
Chronic non-healing ulcer is a common problem met in clinical practice and represents a burden to the patients. Chronic ulcer lacks growth factors (GFs) to promote the healing process and is frequently followed by superadded infections. Ordinary technique such as wound debridement and regular dressings cannot provide adequate results as these techniques cannot provide the necessary GFs. Platelet-rich plasma (PRP) helps wound healing by releasing various types of GFs.

The aim: to evaluate and compare the efficacy of PRP dressing versus traditional dressings in the treatment of chronic non-healing leg and foot ulcers of different etiology as regard cost of overall treatment and effectiveness (reduction of the size of the ulcer and safety of the technique).

Methods

This prospective study was performed on inpatients and outpatients in general surgery department, Zagazig university hospital from June 2017 to January 2019. Patients were divided randomly into two groups: group A received PRP dressing (N=22, 50%) and group B received conventional ordinary dressing (N=22, 50%).The mean follow-up period was 3 months after the last dressing. Patients treated with PRP at once-weekly interval for a maximum of 12 dressings while patients with ordinary dressings may need one dressing every other day for a maximum of 12 weeks. The reduction in the size of the ulcers (area and volume) in both groups was assessed using centimeter scale and Digital photographs before and after each session and during follow up period.

Keywords: Platelet-rich plasma, ulcers, non-healing, ordinary dressing.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old,
* males and non-pregnant females,
* hemoglobin (> 10 gm. /dL),
* post-prandial blood sugar ≤ 140 mg% if diabetic,
* Wounds free of infection (sterile swab) or necrosis.

Exclusion Criteria:

* malignant ulcer(by biopsy),
* pus discharge/slough,
* ulcer with exposed tendons/ligaments/bone,
* ischemic ulcer (by duplex U/S),
* non-compliant patients ,
* radiation near to the site of ulcer,
* osteomyelitis of underlying bone (x-ray-bone scan) ,
* steroids therapy ,
* thrombocytopenia(< 150,000/dl)
* patients unfit or refuse blood donation from himself or from others.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
change the ulcer size | 1.8 years
  healing of the ulcer is assessed using centimeter scale before each dressing

CONTACTS AND LOCATIONS:
Overall Officials: tamer A Alnaimy, MD, Study Director — faculty of medicine Zagazig university
Locations (1):
- Tamer Alsaied Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No